CLINICAL TRIAL: NCT01171326
Title: A Randomized, Parallel-group, Double Blind, Clinical Trial, to Assess the Safety and Efficacy of Topically Applied FXFM244 Antibiotic Foam in the Treatment of Impetigo
Brief Title: Study to Evaluate the Safety and Efficacy of Topical Minocycline FXFM244 in Impetigo Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 005-10LND /FX2010-01
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Impetigo
Keywords: topical; minocycline; foam; phase II; impetigo
MeSH Terms: conditions — Impetigo; cyclopia sequence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Minocycline Foam FXFM244 - 4% (Experimental): Minocycline Foam FXFM244 - 4%
  Interventions: Drug: Topical Minocycline Foam FXFM244
- Topical Minocycline Foam FXFM244 - 1% (Experimental): Minocycline Foam FXFM244 - 1%
  Interventions: Drug: Topical Minocycline Foam FXFM244

INTERVENTIONS:
Drug: Topical Minocycline Foam FXFM244 — FXFM244 - 1%, FXFM244 - 4% to be applied twice daily during 7 days

SUMMARY:
Impetigo is a common, highly infectious skin disease caused by bacterial infection and characterized by crusting skin lesions. It is most common in children, particularly children in unhealthy living conditions. In adults, it may follow other skin disorders. Impetigo is caused primarily by the bacteria Streptococcus pyogenes and/or Staphylococcus aureus, which can also be isolated from impetigo lesions.

This is a pilot phase II study to evaluate the tolerability and safety and to monitor the clinical efficacy of Topical Minocycline Foam FXFM244 in impetigo patients.

DETAILED DESCRIPTION:
A randomized, parallel-group, double (Investigator, patient) blind, comparative dose range finding clinical trial.

The study will involve two treatment groups. Eligible patients will be randomized to receive either FXFM244 - 1%, FXFM244 - 4% , in a blinded fashion. Patients will be treated twice daily for 7 days. Following the screening period and baseline visit, study subjects will return at days 3, 7 and 14. At each visit, patients will be evaluated via lesion count, global assessment tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of pure impetigo, impetigo contagiosa, or uncomplicated blistering impetigo
* Patients 2 years of age or older, and in general good health
* Patients with no less than two lesions and no more than seven lesions, area 0.5x0.5cm.
* No known medical conditions that, in the Investigator's opinion could interfere with study participation
* Patient / Patient's guardian (in the case of children) willing and able to comply with all requirement of the protocol
* Patient / Patient's guardian willing and able to give written informed consent prior to participation in the study

Exclusion Criteria:

* Presence of skin diseases at or near the investigational area
* Immunosuppressed state or other serious systemic disease
* Signs and/or symptoms of systemic infection
* Presence of skin infection/disorder not amenable to topical antibacterial treatment only
* Presence of secondarily-infected animal/human bite
* Presence of secondarily infected burn wound
* Topical or systemic use of medicinal or other products before or during the study (oral or topical antibiotics, oral or topical corticosteroids and immuno modulators); or other drugs, which in the Investigators opinion could confound the evaluation of the effect of the study drugs
* Known or suspected hypersensitivity to Minocycline or any of the excipients in the study medication
* Participation in any other investigational drug study or use of (an) investigational drug(s) within the 30 days or 5 half-lives (whichever is longer) prior to randomization
* Patients previously enrolled/randomized in this study
* Use of another investigational drug within 30 days prior to entry into this study.
* Pregnant or lactating women.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Decrease in lesion count | 7 days

SECONDARY OUTCOMES:
The severity of the overall impetigo condition will be measured at baseline and at all follow-up visits. The severity will be assessed and graded based on the scales for Investigator's Global Assessment and bacteriological testing. | Days 3, 7 and 14

CONTACTS AND LOCATIONS:
Locations (1):
- Lev Yasmin Clinic, Netanya, Israel